CLINICAL TRIAL: NCT05585021
Title: A Clinical Study on The Effect of Probiotic Compound Powder (WONDERLAB) on The Immunity Improvement of Preschool Children (RCT)
Brief Title: Clinical Study on the Effect of Probiotic Compound Powder on the Immunity Improvement of Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Precision Health Food Technology Co. Ltd., (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22-SM-08-WL-001
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Immunity
Keywords: Rotavirus; Upper respiratory tract infection; Bristol scoring method
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: The community hospital will recruit 140 preschool children, aged 5 to 6 years old, according to the inclusion and exclusion criteria, and randomly assigned them to 2 groups. 70 subjects in the placebo group and 70 in the experimental product group.
  First entered a one-week washout period, and then entered a 25-week clinical intervention, and finally ensured that 100 volunteers completed the whole study, and the withdrawal rate was about 28%.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wonderlab Kids instant probiotics (Experimental): Wonderlab Kids instant probiotics (hawthorn flavor) (4 strains, 20 billion CFU/bottle) 2g/bottle
  Interventions: Dietary Supplement: Wonderlab Kids instant probiotics
- Instant probiotic placebo (Placebo Comparator): Instant probiotic placebo (ET) 2g/bottle
  Interventions: Dietary Supplement: Instant probiotic placebo

INTERVENTIONS:
Dietary Supplement: Wonderlab Kids instant probiotics — During study intervention, subjects are required to take the randomly assigned product based on the randomization list.
  Taking assigned product directly or mix it with milk/water/other liquids below 37 ℃, take it half an hour after meal.1 bottle a day. Lasting for 24 weeks intervention period.
  Arms: Wonderlab Kids instant probiotics
Dietary Supplement: Instant probiotic placebo — Subjects are required to take the randomly assigned Instant probiotic placebo based on the randomization list.
  Taking assigned product directly or mix it with milk/water/other liquids below 37 ℃, half an hour after meal.
  1 bottle a day. Lasting for 24 weeks intervention period.
  Arms: Instant probiotic placebo

SUMMARY:
This is a randomized controlled trial, to evaluate the effect of WONDERLAB Probiotic Compound Powder on improving immunity of preschool children

DETAILED DESCRIPTION:
The community hospital will recruit 140 preschool children, aged 5 to 6 years old, according to the inclusion and exclusion criteria, and randomly assigned them to 2 groups. 70 subjects in the placebo group and 70 in the experimental product group.

First entered a one-week washout period, and then entered a 25-week clinical intervention, and finally ensured that 100 volunteers completed the whole study, and the withdrawal rate was about 28%.

ELIGIBILITY:
Inclusion Criteria:

* Preschool children, male or female, 5 to 6 years old;
* Those with weak constitution and easy to get sick:

One of them can be satisfied:

AGet cold ≥ 3 times a year B Bronchitis or pneumonia ≥2 times per year C Rotavirus diarrhea ≥1 time per year

* During the trial, participants agree not to take any drugs, supplements, or other dairy products containing probiotics;
* During the trial, participants agree not to take any other prebiotic/bacterial drugs, supplements, or dairy products including yogurt drinks;
* Willing to refrain from participating in other interventional clinical studies during the trial period;
* Be able to fully understand the nature, purpose, benefits and possible risks and side effects of the research;
* Willing to obey all test requirements and procedures;
* Informed consent signed by parents or legal guardians.

Exclusion Criteria:

* Subject who is in the treatment of gastrointestinal diseases;
* Subject who has lactose intolerance;
* The subjects are currently suffering from other organic diseases that affect intestinal function, such as history of gastrointestinal resection, colonic or rectal cancer, inflammatory bowel disease, diabetes, hyperthyroidism or hypothyroidism, Hirschsprung's disease, scleroderma, anorexia nervosa, etc.;
* Subjects have any of the following medical histories or clinically diagnosed diseases that may affect the evaluation of the test effect: obvious gastrointestinal dysfunction, liver, kidney, endocrine, blood, respiratory and cardiovascular diseases;
* According to the judgment of the researchers, frequent use of drugs that may affect gastrointestinal function or the immune system;
* Subjects who took laxatives or other digestive aids 2 weeks before the start of the study;
* Consumed dairy products or other foods containing prebiotics/bacteria within 10 days before the start of the study;
* PI believes that volunteers cannot fully cooperate with the trial arrangement.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Rotavirus diarrhea Testing at baseline | baseline(day 0)
  Records of sick leave days, medical visits and hospitalization days due to rotavirus infection within past 12 month
Rotavirus diarrhea Testing at endpoint | endpoint( day 168)
  Records of sick leave days, medical visits and hospitalization days due to rotavirus infection within past 168 days
Infection of the upper respiratory tract at baseline | baseline(day 0)
  Drug records of upper respiratory tract infection within past 12 months.
Infection of the upper respiratory tract at endpoint | endpoint ( day 168)
  Drug records of upper respiratory tract infection within past 168 days.

SECONDARY OUTCOMES:
Bristol Stool Chart | baseline(day 0)/interim ( day 84)/endpoint( day 168)/recession period( day 175)
  To evaluate samples of human feces based on the shape and consistency of the stool.
Faeces | baseline(day 0)/interim ( day 84)/endpoint( day 168)/recession period( day 175)
  sIgA 、16sRNA、SCFA、Fecal calprotectin
Saliva | baseline(day 0)/interim ( day 84)/endpoint( day 168)/recession period( day 175)
  sIgA testing
Pittsburgh sleep quality index | baseline(day 0)/interim ( day 84)/endpoint( day 168)
  18 items comprise 7 components, each of which is scored according to o~3 grade. The cumulative score of each component is the total score of PSQI, with a total score range of 0~2l. The higher the score, the worse the sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyang Sheng, MD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Wenan Wang, Jinhua, Zhejiang, China